CLINICAL TRIAL: NCT04023604
Title: Does Antimicrobial-free Production of Beef Cattle Reduce Foodborne Transmission of Resistant Bacteria to Human Consumers?
Brief Title: Antimicrobial-free Production of Beef Cattle's Affect on Gut Microbiome
Acronym: S54
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Colorado State University (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1905022180
Record Dates: First submitted 2019-06-28; First posted 2019-07-17 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Diet Modification
Keywords: antibiotics; gut microbiome; antimicrobial resistance; beef
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: This is a 16-week randomized, cross-over, controlled, blinded study. During weeks 2 and 9, participants usual, unrestricted dietary intakes will be assessed. At week 3 the participants will be randomized and assigned to consume either the controlled U.S. Healthy Eating Pattern with beef produced in conventional systems or to an identical controlled U.S. Healthy Eating Patter with beef produced in RWA (raised without antibiotics) systems. Week 10 will be the second 3- week long dietary intervention period. A total of 14 stool samples will be collected during the study (two after baseline, washout 1 and washout 2, and 4 during the two dietary interventions). Two fasting state serum samples and a psychological questionnaire will be collected during study weeks 2, 5, 9, and 12.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled diet with beef raised without antibiotics (Active Comparator): Subjects will be randomized and assigned to consume the U.S. Healthy Diet Diets with beef produced in RWA (raised without antibiotics) systems for three weeks.
  Interventions: Other: Controlled diet with beef raised without antibiotics
- Controlled diet with beef produced in conventional systems (Experimental): Subjects will be randomized and assigned to consume the U.S. Healthy Diet Diets with beef produced in conventional systems for three weeks.
  Interventions: Other: Controlled diet with beef produced in conventional systems

INTERVENTIONS:
Other: Controlled diet with beef raised without antibiotics — The controlled diet with beef raised without antibiotics will follow the Dietary Guidelines for American's recommendations. All foods and beverages will be provided during intervention to achieve the desired eating pattern. Beef included in this diet were raised without antibiotics.
  Arms: Controlled diet with beef raised without antibiotics
Other: Controlled diet with beef produced in conventional systems — The controlled diet with beef raised without antibiotics will follow the Dietary Guidelines for American's recommendations. All foods and beverages will be provided during intervention to achieve the desired eating pattern. Beef included in this diet were raised with antibiotics.
  Arms: Controlled diet with beef produced in conventional systems

SUMMARY:
The primary purpose of this study is to assess whether consuming foods from animals raised with antimicrobial medications influences gut health in adults between the ages of 21-69 years old. Antimicrobial medications are commonly used to help animals avoid infections while growing.

DETAILED DESCRIPTION:
The researchers plan to investigate differences in the resistome (i.e., populations of antimicrobial resistance genes) and microbiome (populations of bacteria) in feces obtained from people when they consume diets containing beef derived from cattle raised conventionally (i.e. using antimicrobial drugs(AMDs)) vs. those produced in raised without antibiotics (RWA) systems. In addition, the researchers will investigate whether specific antimicrobial resistant (AMR) genes are transmitted from food to people.

The hypothesis is that beef is not a significant source of resistant bacteria, and there is no difference in the likelihood of gut colonization with resistant bacteria in people eating beef derived from cattle raised conventionally (i.e. using AMDs) vs. those eating beef produced in RWA systems.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 21-69 years old;
* BMI 22.0-34.9 kg/m2;
* Fasting serum total cholesterol <240 mg/dL, low-density lipoprotein cholesterol <160 mg/dL, triglycerides <400 mg/dL, and glucose <110 mg/dL;
* Systolic/diastolic blood pressure <140/90 mmHg;
* Body weight stable (± 4 kg in previous 3 mo);
* Medication use stable for 6 months prior and not using medications or supplements known to impact gut function;
* No use of topical, oral or parenteral antibiotic medications in previous 6 months.
* Non-smoking;
* Physical activity regimen stable for 3 months prior;
* Not drinking more than 2 alcoholic drinks per day;
* No history of gastrointestinal disorders, surgeries or cancers;
* Non-pregnant and not lactating
* No acute illness and non-diabetic;
* Willing and able to consume the prescribed diets that may include meat, dairy and gluten-containing foods and beverages.

Exclusion Criteria:

* Male or female, < 20 or >70 years old;
* BMI < 21.9- >35 kg/m2;
* Fasting serum total cholesterol >240 mg/dL, low-density lipoprotein cholesterol >160 mg/dL, triglycerides >400 mg/dL, and glucose >110 mg/dL;
* Systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg;
* Body weight stable for < 3 months prior (±3 kg);
* Stable physical activity regimen < 3 months prior;
* Medication use unstable for 6 months prior and using medications or supplements known to impact gut function;
* Smoking;
* Drinking more than 2 alcoholic drinks per day;
* Diabetic;
* A history of gastrointestinal disorders, GI surgeries or GI cancers;
* Pregnant or lactating

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Differences in the resistome and microbiome | 2 years
  The resistome and microbiome of rinsates will be obtained from dietary components, and feces collected from the particpants. Researchers will sequence all of the published AMR genes. Microbiome data will be obtained from 16s rRNA gene sequencing to produce amplicons of the V4 region of 16S rRNA genes. Statistical analyses will be conducted of microbial features to assess whether microbial/resistome communities diverge between the two groups. Additionally, foodborne transmission of AMR genes with discriminatory SNP("DNA fingerprints") profiles will be investigated through the food chain into dietary trial participants to identify highly discriminatory patterns in individual genes, or discriminatory profiles in gene sets. Hypothesis: beef is not a significant source of resistant bacteria and there is no difference in the likelihood of gut colonization with resistant bacteria in people eating beef derived from cattle raised conventionally vs beef produced in RWA systems

SECONDARY OUTCOMES:
Level of fasting blood pressure | 2 years
  The hypothesis is that there is no difference in blood pressure in people eating beef derived from cattle raised conventionally vs. those eating beef produced in RWA systems.
Level of fasting serum insulin | 2 years
  The hypothesis is that there is no difference in fasting serum insulin in people eating beef derived from cattle raised conventionally vs. those eating beef produced in RWA systems.
Level of fasting serum glucose | 2 years
  The hypothesis is that there is no difference in fasting serum glucose in people eating beef derived from cattle raised conventionally vs. those eating beef produced in RWA systems.
Size of lipoprotein particle | 2 years
  The hypothesis is that there is no difference in lipoprotein particle size in people eating beef derived from cattle raised conventionally vs. those eating beef produced in RWA systems

OTHER OUTCOMES:
Questionnaire score of mood and health and well being | 2 years
  The POMS (Profile of Mood States) Questionnaire is a psychological rating scale to assess distinct mood states. There is a total of 35 questions using a five point scale ranging from "not at all" to "extremely" indicating the range of mood swings over a period of time.
  The Optum SF-36v2 (Short Form 36 question Version 2) Health Survey measures the functional health and wellbeing of a participant. SF-36v2 consists of eight scaled scores which are the weighted sums of the questions in their section. Each scale is transformed into a 0-100 scales, with the assumption that each questions carries equal weight (the lower the score the more disability, the higher the score the less disability).
  The hypothesis is that there is no difference in mood and health and wellbeing in people eating beef derived from cattle raised conventionally vs. those eating beef produced in RWA systems.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, PhD, Principal Investigator — Purdue University
Locations (1):
- Dept. Foods and Nutrition, Purdue University, West Lafayette, Indiana, United States